CLINICAL TRIAL: NCT01138735
Title: A Multi-center, Randomized, Vehicle-controlled, Double-blind, Study to Evaluate the Safety and Efficacy of Epiduo® (Adapalene and Benzoyl Peroxide) Gel 0.1%/2.5% Administered Once Daily for the Treatment of Subjects 9 to 11 Years of Age With Acne Vulgaris
Brief Title: Epiduo Pediatric Acne Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18155
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Results first posted 2013-03-26 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2013-04

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination; Adapalene; Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- adapalene/benzoyl peroxide (Active Comparator): Epiduo® (adapalene and benzoyl peroxide) Gel 0.1%/2.5% applied topically once daily for 12 weeks
  Interventions: Drug: adapalene/benzoyl peroxide
- Topical Gel Vehicle (Placebo Comparator): Topical Gel Vehicle applied topically once daily for 12 weeks
  Interventions: Drug: Topical Gel Vehicle

INTERVENTIONS:
Drug: adapalene/benzoyl peroxide — daily topical application for 12 weeks
  Other Names: Epiduo® (adapalene and benzoyl peroxide) Gel 0.1%/2.5%
  Arms: adapalene/benzoyl peroxide
Drug: Topical Gel Vehicle — daily topical application for 12 weeks
  Arms: Topical Gel Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Epiduo® (adapalene and benzoyl peroxide) Gel 0.1%/2.5% administered once daily for up to 12 weeks in subjects 9 to 11 years of age with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acne vulgaris with facial involvement
* Score of 3 (moderate) on the Investigator's Global Assessment (IGA) scale
* A minimum of 20 but not more than 100 total lesions (Noninflammatory and/or Inflammatory) on the face (including the nose) at Baseline

Exclusion Criteria:

* Acne nodule or acne cyst
* Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), or severe acne requiring systemic treatment
* Underlying diseases and/or dermatologic conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments
* Use of prohibited medications prior to the study and/or are unwilling to refrain from such use during the study

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D; Lorne Albrecht, MD, Principal Investigator — Guildford Dermatology Specialists; Zoe Draelos, MD, Principal Investigator — Zoe Draelos, MD; Lawrence Eichenfield, MD, Principal Investigator — Childrens Hospital and Health Center Division of Pediatric and Adolescent Dermatology; Boni Elewski, MD, Principal Investigator — UAB Dermatology Clinical Research; Alan Fleischer, MD, Principal Investigator — Department of Dermatology Wake Forest University Health Sciences; Francisco Flores, MD, Principal Investigator — FXM Research Miramar; Joseph Fowler, MD, Principal Investigator — Dermatology Specialists Research; Robert Haber, MD, Principal Investigator — Haber Dermatology Clinical Research Center; Adelaide Hebert, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Michael Heffernan, MD, Principal Investigator — Central Dermatology, PC; David Kaplan, MD, Principal Investigator — Adult & Pediatric Dermatology; Steven Kempers, MD, Principal Investigator — Minnesota Clinical Study Center A Division of Associated Skin Care Specialist, PA; Rodion Kunynetz, MD, Principal Investigator — Ultranova Skincare; Ian Landells, MD, Principal Investigator — Nexus Clinical Research; Charles Lynde, MD, Principal Investigator — Lynderm Research Inc.; Russell Mader, MD, Principal Investigator — Dermatology Associates of Kingsport, PC; Lew Andrew Rosoph, MD, Principal Investigator — North Bay Dermatology Centre; Joel Schlessenger, MD, Principal Investigator — Skin Specialists, PC; Michael Spigarelli, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Linda Stein Gold, MD, Principal Investigator — Henry Ford Health Systems - Department of Dermatology; Jeffrey Sugarman, MD, Principal Investigator — Redwood Family Dermatology; William Werschler, MD, Principal Investigator — Premier Clinical Research; Patricia Westmoreland, MD, Principal Investigator — Palmetto Clinical Trial Services, LLC; Andrea Zaenglein, MD, Principal Investigator — Penn State Milton S. Hershey Medical Center - Penn State College of Medicine; George Murakawa, MD, Principal Investigator — Dermcenter PC; Somerset Skin Centre
Locations (25):
- United States (20):
  - UAB Dermatology Clinical Research, Birmingham, Alabama
  - Children's Hospital and Health Center Division of Pediatric and Adolescent Dermatology, San Diego, California
  - Redwood Family Dermatology, Santa Rosa, California
  - FXM Research Miramar, Miramar, Florida
  - Adult & Pediatric Dermatology, Overland Park, Kansas
  - Dermatology Specialists Research, Louisville, Kentucky
  - Henry Ford Health Systems Department of Dermatology, Detroit, Michigan
  - Dermcenter PC - Somerset Skin Centre, Troy, Michigan
  - Minnesota Clinical Study Center A Division of Associated Skin Care Specialists, PA, Fridley, Minnesota
  - Central Dermatology PC, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Zoe Draelos, MD, High Point, North Carolina
  - Department of Dermatology - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cininnati Children's Hospital, Cincinnati, Ohio
  - Haber Dermatology Clinical Research Center, South Euclid, Ohio
  - Penn State Milton S. Hershey Medical Center - Penn State College of Medicine, Hershey, Pennsylvania
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Dermatology Associates of Kingsport, PC, Kingsport, Tennessee
  - The University of Texas Health Sciences Center at Houston, Houston, Texas
  - Premier Clinical Research, Spokane, Washington
- Canada (5):
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Ultranova Skincare, Barrie, Ontario
  - Lynderm Research, Inc, Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adapalene/Benzoyl Peroxide | Topical Gel Vehicle
Started | 142 | 143
Completed | 134 | 126
Not Completed | 8 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene/Benzoyl Peroxide | Topical Gel Vehicle | Total
Number analyzed (Participants) | 142 | 143 | 285
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 142 | 143 | 285
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (0.76) | 10.4 (0.68) | 10.4 (0.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 108 | 217
  Male | 33 | 35 | 68
Region of Enrollment [Number; unit: participants]
  United States | 130 | 129 | 259
  Canada | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Percentage of subjects rated Clear or Almost Clear with at least 2 grades reduction from Baseline on the Investigator's Global Assessment (IGA)
Time Frame: Baseline to Week 12 (Last Observation Carried Forward [LOCF])
Population: Intent to treat (ITT) population, LOCF
Measure: Number; unit: percentage of participant
Arm/Group | Adapalene/Benzoyl Peroxide | Topical Gel Vehicle
Number analyzed (Participants) | 142 | 143
percentage of participant | 47.2 | 15.4
Statistical Analysis 1: Comparison: Adapalene/Benzoyl Peroxide vs Topical Gel Vehicle; null hypothesis: no difference in Success rate in two treatment groups (adapalene/benzoyl peroxide vs Topical Gel Vehicle). power calculation: 90%; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustment for multiplicity is required. The tests will be conducted as two-sided, each at the 0.05 significance level. The trial will be claimed 'positive' if all primary analyses are shown statistically significant at the 0.05 level; Cochran-Mantel-Haenszel(CMH) test stratified by analysis center, using general association statistics

2. Primary Outcome: Change From Baseline in Total Lesion Counts
Time Frame: Baseline to Week 12 (LOCF)
Population: ITT population, LOCF
Measure: Mean (Standard Deviation); unit: lesion count change
Arm/Group | Adapalene/Benzoyl Peroxide | Topical Gel Vehicle
Number analyzed (Participants) | 142 | 143
lesion count change | -27.6 (22.43) | -3.6 (24.44)
Statistical Analysis 1: Comparison: Adapalene/Benzoyl Peroxide vs Topical Gel Vehicle; null hypothesis: no difference in change from baseline in total lesion count in two treatment groups (adapalene/benzoyl peroxide vs Topical Gel Vehicle); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; normality assumption is not met. ANCOVA Model: Ranked Change in Total Lesion Counts = Ranked Baseline Lesion Counts, Analysis Center, Treatment

3. Secondary Outcome: Percent Change in Total Lesion Counts From Baseline
Time Frame: Baseline to Week 12 (LOCF)
Population: ITT Population, LOCF
Measure: Mean (Standard Deviation); unit: percentage of change in lesion count
Arm/Group | Adapalene/Benzoyl Peroxide | Topical Gel Vehicle
Number analyzed (Participants) | 142 | 143
percentage of change in lesion count | -55.5 (38.99) | -9.3 (48.00)
Statistical Analysis 1: Comparison: Adapalene/Benzoyl Peroxide vs Topical Gel Vehicle; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH test with row mean difference statistic using relative to an identified distribution(RIDIT) score, controlling for analysis center

4. Secondary Outcome: Change in Inflammatory Lesion Counts From Baseline
Time Frame: Baseline to Week 12 (LOCF)
Population: ITT Population, LOCF
Measure: Mean (Standard Deviation); unit: lesion count change
Arm/Group | Adapalene/Benzoyl Peroxide | Topical Gel Vehicle
Number analyzed (Participants) | 142 | 143
lesion count change | -7.4 (12.46) | -0.7 (12.46)
Statistical Analysis 1: Comparison: Adapalene/Benzoyl Peroxide vs Topical Gel Vehicle; Test type: Superiority or Other; p < 0.001, ANCOVA; Ranked Change in Inflammatory Lesion Counts = Ranked Baseline Inflammatory Lesion Counts, Analysis Center, Treatment

ADVERSE EVENTS:
Arm/Group | Adapalene/Benzoyl Peroxide | Topical Gel Vehicle
Serious Adverse Events (participants affected / at risk) | 0/142 | 1/143
Other Adverse Events (participants affected / at risk) | 37/142 | 18/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene/Benzoyl Peroxide (N=142) | Topical Gel Vehicle (N=143)
RIGHT FRONTAL ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — occurred on Day 2, resolved on Day 29 and the subject completed the study as planned.Severe, nonrelated Adverse Events (AE), Inpatient hospitalization.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adapalene/Benzoyl Peroxide (N=142) | Topical Gel Vehicle (N=143)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 14 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 8 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 5
Nasopharyngitis (Infections and infestations) | 8 | 13

LIMITATIONS AND CAVEATS:
LOCF data were used for primary efficacy and secondary efficacy data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other